CLINICAL TRIAL: NCT04725682
Title: A Single Dose, Open-Label, Randomized, Four-Way Crossover, Fully Replicate, Bioequivalence Study of Generic Tacrolimus and Prograf® Capsules in Healthy Volunteers Under Fasting Conditions
Brief Title: Bioequivalence Study of Tacrolimus in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Food and Drug Administration (FDA) (U.S. Federal Agency)
Collaborators: BioPharma Services Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Protocol 2521
Record Dates: First submitted 2021-01-15; First posted 2021-01-27 (Actual); Results first posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Healthy Volunteers
Keywords: generic drug; tacrolimus; bioequivalence; reference listed drug; fasting condition
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Intervention Model Description: a single-dose, randomized, open-label, four-period, two-sequence, two- treatment, single-center, crossover, bioequivalence study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sequence 1 (TRTR) (Active Comparator): Each subject is scheduled to receive each treatment twice by the end of the study in the order of TRTR.
  Treatment T (Test): 1 × 1mg Test tacrolimus capsules (Applicant holder: Accord Healthcare, Inc.); Treatment R (Reference): 1 × 1mg RLD tacrolimus capsules
  Interventions: Drug: Tacrolimus
- Sequence 2 (RTRT) (Active Comparator): Each subject is scheduled to receive each treatment twice by the end of the study in the order of RTRT.
  Treatment T (Test): 1 × 1mg Test tacrolimus capsules (Applicant holder: Accord Healthcare, Inc.); Treatment R (Reference): 1 × 1mg RLD capsules
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Tacrolimus — a single dose of 1 mg capsule per period

SUMMARY:
This is an in-vivo study to investigate the bioequivalence of generic tacrolimus and its reference listed drug (RLD). The objective of this study is to investigate the bioequivalence of generic Tacrolimus and RLD in healthy male and non-pregnant, non-lactating female volunteers under fasting conditions. The outcome of this study will help further understanding about pharmacokinetic (PK) performance of tacrolimus in a healthy volunteer population and improve review standards for bioequivalence of narrow therapeutic index (NTI) drugs.

DETAILED DESCRIPTION:
This is a single-dose, randomized, open-label, fully replicate crossover, four-period, two- treatment, two-sequence, bioequivalence study to investigate the bioequivalence of generic tacrolimus and its reference listed drug (RLD).

Tacrolimus, a calcineurin inhibitor (CNI), has been widely used in solid organ and bone marrow transplants for more than two decades. Calcineurin, a calcium-dependent phosphatase, is instrumental for signal transduction for activation of T cell and B cell, which in turn cause production of autoinflammatory cytokines such as such as interleukin 2 (IL- 2), tumor necrosis factor-alpha (TNF-α), and interferon-gamma (IFN-γ). CNIs prevents the dephosphorylation and translocation of various factors such as the nuclear factor of activated T-cells (NF-AT), and nuclear factor kappa-light-chain enhancer of activated B-cells (NF-κB), thereby inhibiting the signal transduction responsible for growth and proliferation of activated T cells and expression of autoinflammatory cytokines. This mechanism of action results in immunosuppression and prevents organ rejection.

However, therapeutic drug monitoring is required for tacrolimus since the range between tacrolimus therapeutic and toxic tacrolimus whole blood concentrations is narrow and some toxicities are serious and/or irreversible. The objective of this study is to investigate the bioequivalence of generic Tacrolimus and RLD in healthy male and non-pregnant, non-lactating female volunteers under fasting conditions.

The outcome of this study will help further understanding about pharmacokinetic (PK) performance of tacrolimus in a healthy volunteer population and improve review standards for bioequivalence of narrow therapeutic index (NTI) drugs.

ELIGIBILITY:
Inclusion Criteria:

1. Males and female volunteers, 18 -59 years of age (inclusive).
2. BMI that is within 18.5-33.0 kg/m², inclusive.
3. Healthy, according to medical history, ECG, vital signs, laboratory results and physical examination as determined by the PI/Sub-Investigator.
4. Capable of giving written informed consent prior to receiving any study medication.
5. Availability to volunteer for the entire study duration and willing to adhere to all protocol requirements.
6. Smokers: Capable of refraining from smoking for the duration of the confinement.
7. Female subjects must be non-pregnant, non-lactating and fulfill at least one of the following:

   * Be surgically sterile for a minimum of 6 months
   * Post-menopausal for a minimum of 12 months; Menopause defined as 12 months of amenorrhea without any other obvious pathological or physiological cause.
   * Agree to avoid pregnancy and use medically acceptable method of contraception from at least 30 days prior to the study until 30 days after the study has ended (last study procedure).

   Medically acceptable methods of contraception include non-hormonal intrauterine device or double barrier method (foam or vaginal spermicidal suppository in conjunction with a male condom, diaphragm with spermicide in conjunction with a male condom). Abstinence as a method of contraception is acceptable if it is in line with the preferred and usual lifestyle of the study participant.

   If a female subject becomes pregnant during participation in the study or within 30 days after she has completed her last tacrolimus administration (whichever was administered last), she must inform BPSUSA staff immediately.
8. Males who are able to father children must agree to use medically acceptable methods of contraception and not to donate sperm during the study and for 30 days after the end of the study.

Medically acceptable methods of contraception include using a condom with a female partner of child-bearing potential who is using: oral contraceptives, hormonal patch, implant or injection, intrauterine device, or diaphragm with spermicide.

If a male subject's partner becomes pregnant during his participation in the study or within 30 days after he has completed his last tacrolimus administration (whichever was administered last), he must inform BPSUSA staff immediately.

Exclusion Criteria:

1. Known history and/or presence of any clinically significant hepatic (e.g., hepatitis, jaundice, hepatic failure, hepatic necrosis, hepatic encephalopathy, biliary tract diseases, cirrhosis), renal/genitourinary (e.g., urethral stricture, any renal impairment), gastrointestinal, cardiovascular (e.g., hypotension including orthostatic hypotension, cor pulmonale, congenital long QT, congestive heart failure, bradyarrhythmias), cerebrovascular, pulmonary (e.g., chronic obstructive pulmonary disease, decreased respiratory reserve, hypoxia, pre-existing respiratory depression), endocrine (e.g., myxedema, hypothyroidism, adrenal cortical insufficiency), immunological, musculoskeletal (e.g., kyphoscoliosis), neurological (e.g., CNS depression or coma, increased cerebrospinal pressure), psychiatric (e.g., psychosis, depression, hallucinations, delirium tremens, suicidal thoughts or behavior), dermatological or hematological (e.g., thrombocytopenic purpura) disease or condition unless determined as not clinically significant by the PI/Sub- Investigator.
2. History or presence of any clinically significant gastrointestinal pathology (e.g., chronic diarrhea, inflammatory bowel disease), unresolved gastrointestinal symptoms (e.g., diarrhea, vomiting), or other conditions known to interfere with the absorption, distribution, metabolism or excretion of the drug experienced within 7 days prior to first tacrolimus administration, as determined by the PI/Sub-Investigator.
3. Systolic blood pressure outside 90-130 mmHg, inclusive, and diastolic blood pressure outside 55-80 mmHg, inclusive, and heart rate between 50-100 bpm, inclusive, unless deemed otherwise by the PI/Sub-Investigator.
4. QTc interval ≥ 440 milliseconds for males and ≥ 460 milliseconds for females, unless deemed otherwise by the PI/Sub-Investigator.
5. Abnormal clinical laboratory values unless values are deemed by the PI/Sub- Investigator as "Not Clinically Significant".
6. Abnormal vital signs (blood pressure [BP], heart rate [HR], respiratory rate [RR], pulse oximetry and temperature) measurements, unless deemed otherwise by the PI/Sub-Investigator.
7. Presence of any clinically significant illness within 30 days prior to first dosing, as determined by the PI/Sub-Investigator.
8. Presence of any significant physical or organ abnormality as determined by the PI/Sub-Investigator.
9. A positive test result for any of the following: HIV, Hepatitis B surface antigen, Hepatitis C, drugs of abuse (marijuana, amphetamines, barbiturates, cocaine, opiates, phencyclidine and benzodiazepines), and alcohol test. Positive serum or urine pregnancy test for female subjects.
10. Known history or presence of:

    * Alcohol abuse or dependence within one year prior to first study drug administration;
    * Drug abuse or dependence;
    * Hypersensitivity or idiosyncratic reaction to tacrolimus, its excipients, and/or related substances;
    * Lymphoma and other malignancies (particularly of the skin);
    * Bacterial, viral, fungal and protozoal infections (e.g., polyoma virus- associated nephropathy [PVAN] due to BK virus infection, JC virus associated progressive multifocal leukoencephalopathy [PML], Epstein Barr Virus (EBC) associated Post transplant lymphoproliferative disorder [PTLD], cytomegalovirus (CMV) infections associated CMV viremia and CMV disease);
    * Tuberculosis;
    * Posterior reversible encephalopathy syndrome (PRES);
    * Pure red cell aplasia (PRCA);
    * Gastrointestinal perforation;
    * Hyperkalemia;
    * Hypertension;
    * Lactose intolerance, galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption;
    * Food allergies and/or presence of any dietary restrictions unless deemed by the PI/Sub-I as "Not Clinically Significant".
    * Severe allergic reactions (e.g. anaphylactic reactions, angioedema).
11. History of intolerance to and/or difficulty with blood sampling through venipuncture.
12. Abnormal diet patterns (for any reason) during the four weeks preceding the study, including fasting, high protein diets, vegan, etc.
13. Individuals who have donated, in the days prior to first tacrolimus administration:

    * 50-499 mL of blood in the previous 30 days;
    * 500 mL or more or double red blood cell ("Power red") donation in the previous 56 days.
14. Donation of plasma by plasmapheresis within 7 days prior to first tacrolimus administration.
15. Hemoglobin level of 12.0 g/dL or lower.
16. Individuals who have participated in another clinical trial or who received an investigational drug within 30 days prior to first tacrolimus administration.
17. Not being able to fast for at least 14 hours.
18. Consumption of food or beverages containing grapefruit and/or pomelo within 3 days prior to first study drug administration.
19. Consumption of food or beverages containing caffeine/methylxanthines, poppy seeds and/or alcohol within 48 hours before dosing in each study period.
20. Use of any prescription medication within 14 days prior to first tacrolimus administration (except for allowed contraceptive products).
21. Use of any over-the-counter medications (including low-dose aspirin, oral multivitamins, allergy medications, herbal and/or dietary supplements) within 14 days prior to first tacrolimus administration (except for spermicidal/barrier contraceptive products).
22. Use of any enzyme-modifying drugs and/or other products, including inhibitors of cytochrome P450 (CYP) enzymes such as antifungals (e.g., ketoconazole, itraconazole, fluconazole, voriconazole, posaconazole, clotrimazole), macrolide antibiotics (e.g., erythromycin, clarithromycin, josamycin), protease inhibitors (e.g., ritonavir, telaprevir [IncivekTM], boceprevir [VictrelisTM], nelfinavir [Viracept®], saquinavir), calcium channel blockers (e.g., verapamil, diltiazem, nifedipine, nicardipine), nucleotide reverse transcriptase inhibitors (e.g., tenofovir), gastric acid, suppressors/neturalizers (e.g., lansoprazole, omeprazole, cimetidine, cisapride, magnesium-aluminum hydroxide antacids), bromocriptine, cortisone, dapsone, ergotamine, gestodene, lidocaine, mephenytoin, miconazole, midazolam, nilvadipine, quinidine, tamoxifen, and triacetyl- oleandomycin and inducers of CYP enzymes such as anti-myobacterials (e.g., rifampin, rifabutin), antifungal agent (e.g., caspofungin), anticonvulsants (e.g. phenytoin, carbamazepine, phenobarbital), corticosteroids (e.g. prednisolone or methylprednisolone), metamizole, isoniazid and products containing St. John's Wort in the previous 30 days before first study drug administration.
23. Use of medicines such as, mycophenolic acid (MPA) products, aminoglycosides, gyrase inhibitors, vancomycin, cotrimoxazole, NSAIDs, oral anticoagulants, or oral antidiabetics, ganciclovir, acyclovir, amphotericin B, ibuprofen, cisplatin, potassium supplements, potassium- sparing diuretics (e.g., amiloride, triamterene or spironolactone), ACE inhibitors (for example, benazepril, enalapril, quinapril), statins (for example, atorvastatin, fluvastatin, simvastatin), angiotensin receptor blockers (for example, irbesartan, valsartan, azilsartan), nefazodone, metoclopramide, danazol, and herbal products containing Schisandra sphenanthera extracts should be avoided during treatment with tacrolimus in the previous 30 days before first study drug administration.
24. Use of any QT prolonging drugs (e.g., citalopram, chlorpromazine, haloperidol, methadone), amiodarone [CordaroneTM, NexteroneTM, PaceroneTM], immunosuppressive or immunomodulating therapies (e.g. sirolimus [Rapamune®], cyclosporins [Gengraf®, Neoral®, and Sandimune®], antilymphocytic antibodies [e.g., basiliximab, daclizumab]) should be avoided during treatment with tacrolimus in the previous 30 days before first study drug administration.
25. Individuals having undergone any major surgery within 6 months prior to the start of the study, unless deemed otherwise by PI/Sub-Investigator.
26. Does not agree, to refrain from driving or operating heavy machinery if feeling dizzy or drowsy following tacrolimus administration until full mental alertness is regained.
27. Does not have an ability to fast for at least 14 hours.
28. Recent history (within 8 weeks prior to screening) of travel to or emigration from any country with high incidence of tuberculosis.
29. Temperature at visit is ≥ 100.4 F° (38.0°C).
30. Test positive for SARS-CoV-2 by locally available, verified test.
31. Have had common symptoms of COVID-19 currently or in the past 14 days as documented in the COVID-19 screening questionnaire and symptom checklist
32. Have had an exposure to suspected or confirmed cases of COVID-19 in the past two weeks as documented in the COVID-19 screening questionnaire
33. Recent live attenuated vaccine1 recipients in the past month.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2021-05-14 (Actual); Study Completion 2021-06-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Artan Markollari, MD, Principal Investigator — BioPharma Services Inc.
Locations (1):
- BioPharma Services USA, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Plan is to make the deidentified, participant data that underlie the results reported in a publication available to researchers who provide a methodologically sound proposal. In addition, the protocol will be made available online at this registry.
Supporting Information: Study Protocol
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal.

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence 1 (TRTR): Each subject is scheduled to receive each treatment twice by the end of the study in the order of TRTR.
  Treatment T (Test): 1 × 1mg Test tacrolimus capsules Treatment R (Reference): 1 × 1mg RLD tacrolimus capsules
  Tacrolimus: a single dose of 1 mg capsule per period
- Sequence 2 (RTRT): Each subject is scheduled to receive each treatment twice by the end of the study in the order of RTRT.
  Treatment T (Test): 1 × 1mg Test tacrolimus capsules Treatment R (Reference): 1 × 1mg RLD capsules
  Tacrolimus: a single dose of 1 mg capsule per period
Period: Overall Study
Arm/Group | Sequence 1 (TRTR) | Sequence 2 (RTRT)
Started | 33 | 34
Completed | 23 | 26
Not Completed | 10 | 8
Not completed — Withdrawal by Subject | 7 | 5
Not completed — Failed to comply with the requirements | 2 | 1
Not completed — Adverse Event | 1 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Participants: This is a crossover study. Participants were randomized to one of the two sequences and were to receive all interventions.
Arm/Group | All Participants
Number analyzed (Participants) | 67
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 67
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 39.0 [24 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 65
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 52
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 67

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration (AUC 72)
Description: Measurement of whole blood tacrolimus prior to dosing and up to 72 hours post-dose
Time Frame: 72 hours
Population: Participants in the PK population with available data.
Measure: Mean (Standard Deviation); unit: pg.h/mL
Groups:
- Tacrolimus (Generic): 1 x 1 mg Tacrolimus capsule (Test)
- Tacrolimus (Brand): 1 x 1 mg Tacrolimus capsule (Reference)
Arm/Group | Tacrolimus (Generic) | Tacrolimus (Brand)
Number analyzed (Participants) | 62 | 61
pg.h/mL | 37434.51 (20086.16) | 33716.80 (19885.62)

2. Primary Outcome: Maximum Plasma Concentration (Cmax)
Description: Measurement of whole blood tacrolimus prior to dosing and up to 144 hours post-dose
Time Frame: 0.25, 0.50, 0.75, 1.00, 1.25, 1.50, 1.75, 2.00, 2.25, 2.50, 2.75, 3.00, 3.50, 4.00, 5.00, 6.00, 8.00, 10.00, 12.00, 16.00, 24.00, 36.00, 48.00, 72.00, 96.00, 120.00, 144.00 hours
Population: Participants in the PK population with available data.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Tacrolimus (Generic) | Tacrolimus (Brand)
Number analyzed (Participants) | 62 | 62
pg/mL | 6780.05 (2830.05) | 4246.68 (2243.37)

3. Secondary Outcome: Time at Maximum Plasma Concentration (Tmax)
Description: Measurement of whole blood tacrolimus prior to dosing and up to 144 hours post-dose
Time Frame: as for outcome 2
Population: Participants in the PK population with available data.
Measure: Median (Full Range); unit: hour
Arm/Group | Tacrolimus (Generic) | Tacrolimus (Brand)
Number analyzed (Participants) | 62 | 62
hour | 1.00 [0.5 to 2.75] | 1.50 [0.75 to 4.03]

4. Secondary Outcome: Area Under the Concentration (AUC Inf)
Description: Time curve from time zero to infinity, calculated as AUCt + Clast/λ, where Clast is the last measurable concentration. Measurement of whole blood tacrolimus prior to dosing and up to 144 hours post-dose.
Time Frame: Estimated using the last measurable concentration (144 hours)
Population: Participants in the PK population with available data.
Measure: Mean (Standard Deviation); unit: pg.h/mL
Arm/Group | Tacrolimus (Generic) | Tacrolimus (Brand)
Number analyzed (Participants) | 61 | 58
pg.h/mL | 45484.38 (25524.52) | 42764.68 (25066.88)

5. Secondary Outcome: Area Under the Concentration (AUC 0-t)
Description: Area under the concentration-time curve from time zero until the last measurable concentration or last sampling time t, whichever occurs first.
Time Frame: To the last measurable concentration or last sampling time t, whichever occurs first. (0 to 144 hours post-dose)
Population: Participants in the PK population with available data.
Measure: Mean (Standard Deviation); unit: pg.h/mL
Arm/Group | Tacrolimus (Generic) | Tacrolimus (Brand)
Number analyzed (Participants) | 61 | 58
pg.h/mL | 41480.11 (24938.47) | 38744.54 (23985.82)

ADVERSE EVENTS:
Time Frame: Approximately 2 months
Description: Safety population included all dosed participants.
Arm/Group | Tacrolimus (Generic) | Tacrolimus (Brand)
All-Cause Mortality (participants affected / at risk) | 0/66 | 1/64
Serious Adverse Events (participants affected / at risk) | 0/66 | 1/64
Other Adverse Events (participants affected / at risk) | 8/66 | 11/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tacrolimus (Generic) (N=66) | Tacrolimus (Brand) (N=64)
Death (General disorders) | 0 (0) | 1 (1) — Unknown cause that occurred during a washout period.
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tacrolimus (Generic) (N=66) | Tacrolimus (Brand) (N=64)
Headache (Nervous system disorders) | 7 | 5
Toothache (Gastrointestinal disorders) | 0 | 2
Vessel puncture site pain (General disorders) | 0 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hypertension (Vascular disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-22): https://cdn.clinicaltrials.gov/large-docs/82/NCT04725682/Prot_SAP_000.pdf